CLINICAL TRIAL: NCT05099536
Title: A Phase I Study of the Safety, Tolerability, Pharmacokinetics Profiles and Preliminary Efficacy of 3D011-08 for Injection Monotherapy in Subjects With Advanced Solid Tumors
Brief Title: 3D011-08 Monotherapy in Subjects With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Company's decision
Sponsor: 3D Medicines (Beijing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: 3D Medicines (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3D011-CN-001
Record Dates: First submitted 2021-10-11; First posted 2021-10-29 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D011-08 (Experimental)
  Interventions: Drug: 3D011-08

INTERVENTIONS:
Drug: 3D011-08 — participants will receive 15mg (starting dose)intravenous drop of 3D011-08,All subjects in each cohort will receive a single dose of 3D011-08 first, followed by a 7-day washout period (i.e. single-dose PK study period). Then, subjects will receive consecutive doses on 1,3,5day of each week (28 days/cycle) until disease progression, death, unacceptable toxicity, or withdraw of informed consent, whichever comes first.Dose of the study medication will be escalated sequentially till the dose limiting toxicity is achieved to determine the recommended part 2 doses (RPTD).

SUMMARY:
The purpose of this study is evaluate the the safety, tolerability, pharmacokinetics profiles, and preliminary efficacy of 3D011-08 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
Detailed Description: This study was initiated on February 24, 2022, at Fudan Cancer Hospital. However, noparticipants were screened or enrolled after the initiation. Due to strategic development adjustments, thecompany terminated the study on September 11. 2023.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic malignant solid tumors(part 1 dose escalation); Histologically confirmed locally advanced or metastatic hepatocellular carcinoma (cohort 1),advanced renal cell carcinoma (cohort 2), and metastatic castration-resistant prostate cancer (cohort 3) for which not amenable to local therapy.(part 2 dose expansion).
2. Cohort 1 and 2: at least one measurable lesion (according to RECIST 1.1 criteria);Cohort 3: at least one measurable or unmeasurable lesion (according to RECIST 1.1 criteria).
3. Subjects must have failed or have been intolerant to established standard therapies, or standard therapies did not exist or were no longer effective for a given tumor type, or in the opinion of the Investigator have been considered ineligible for a particular form of standard therapy on medical grounds(part 1 dose escalation). Cohort 1 (advanced hepatocellular carcinoma)and Cohort 2 (advanced renal cell carcinoma): Subjects had disease progression after received previous first-line of systemic treatment, or subjects are intolerant of or have refused to receive first-line of systemic treatment.

   Cohort 3 (metastatic castration-resistant prostate cancer) : Patients who had failed or had refused prior abiraterone and/or docetaxel chemotherapy.(part 2 dose expansion)
4. ECOG Performance Status ≤ 2(part 1 dose escalation).≤ 1.(part 2 dose expansion)
5. Life expectancy ≥ 12 weeks.
6. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Investigational products or devices in other clinical trials or received antibody drug therapy within 4 weeks before the first dose,or chemotherapy, targeted therapies,or radiotherapy within 2 weeks before the first dose.
2. Participants need to continue using medications known to have a significant risk of causing QTc prolongation or a CYP3A4 strong inhibitor or strong inducer.
3. Participants who have previous toxicity of anti-tumor therapy that has not been returned to level 0 or 1.
4. Participants with diseases at risk of bleeding within 3 months prior to enrollment
5. Participants with concomitant medical conditions requiring anticoagulant therapy at a therapeutic dose
6. History or current condition of uncontrolled cardiovascular disease.
7. Participants with gastrointestinal disease associated with a risk of perforation or fistula formation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of3D011-08 | 24 months
  The maximum tolerated dose as determined in Part 1 of the study will be used as the recommended dose for Part 2.
ORR | 24 Months
  proportion of subjects in cohort 1 and cohort 2 who achieved a confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 as assessed by investigators.
TTP | 24 Months
  time to progression based on the PCWG3 recommendations for assessment of prostate cancer disease progression (CT/MRI, bone scan) as assessed by investigators .

SECONDARY OUTCOMES:
RPTD | 24 months
  RP2D will be determined based on pharmacodynamics or clinical response, as well as the incidence rate and nature of the toxicities observed.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 24 months
Cmax Cmax | 24 months
Css min | 24 months
Tmax | 24 months
AUC0~t、AUC0~∞ | 24 months
Ctrough | 24 months
t1/2 | 24 months
CL | 24 months
Vd | 24 months
ORR | 24 months
  proportion of subjects in part of Dose Escalation who achieved a confirmed complete response (CR) or partial response (PR) based on RECIST v1.1 as assessed by investigators.proportion of subjects in dose expansion cohort 3 who achieved a confirmed complete response (CR) or partial response (PR) based on the PCWG3 recommendations for assessment of prostate cancer disease progression (CT/MRI, bone scan) as assessed by investigators .
Duration of response (DoR) | 24 months
  DoR is defined as the time from the date of first CR or PR based on RECIST v1.1 to the date of first documented progressive disease based on RECIST v1.1 or death, whichever occurs first.part1 Dose Escalation，part 2 dose expansion:Cohort 1 and Cohort 2.
Disease control rate (DCR) | 24 months
  defined as the proportion of subjects who achieve a confirmed complete response (CR) or partial response (PR) or stable disease (SD) based on RECIST v1.1 as assessed by investigators.Proportion of subjects in dose expansion cohort 3 who achieve a confirmed complete response (CR) or partial response (PR) or stable disease (SD) based on the PCWG3 recommendations for assessment of prostate cancer disease progression (CT/MRI, bone scan) as assessed by investigators .
Progression-free survival (PFS) | 24 months
  PFS is defined as the time from the date of first study dose to disease progression based on RECIST v1.1 or death, whichever occurs first. Subjects in dose expansion cohort 3 based on the PCWG3 recommendations for assessment of prostate cancer disease progression (CT/MRI, bone scan) as assessed by investigators .
Permeable surface area of capillary wall(PS) | 24 months
the incremental Area Under Curve (iAUC) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: dingwei Ye, Dr, Principal Investigator — Fudan University; jiang zhang, Dr, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Floor 2, Building 2, 270 Dong 'an Road, Xuhui District, China

IPD SHARING:
Plan to Share IPD: No